CLINICAL TRIAL: NCT03308565
Title: Phase I Clinical Trial of Autologous Adipose Derived Mesenchymal Stem Cells in the Treatment of Paralysis Due to Traumatic Spinal Cord Injury
Brief Title: Adipose Stem Cells for Traumatic Spinal Cord Injury
Acronym: CELLTOP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mohamad Bydon (Other)
Responsible Party: Sponsor-Investigator, Mohamad Bydon, Regulatory Sponsor, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-004621
Record Dates: First submitted 2017-10-09; First posted 2017-10-12 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Spinal Cord Injuries; Paralysis
Keywords: AIS grade A or B
MeSH Terms: conditions — Spinal Cord Injuries; Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase I (Experimental): Patients will receive a single dose of 100 million autologous, adipose derived mesenchymal stem cells. The cells are isolated from patient's adipose tissue and expanded for intrathecal delivery.
  Interventions: Biological: Autologous, Adipose derived Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Autologous, Adipose derived Mesenchymal Stem Cells — The mesenchymal stem cells will be collected and expanded from the subjects adipose tissue.

SUMMARY:
The purpose of this study is to determine if mesenchymal stem cells (MSC) derived from the fat tissue can be safely administered into the cerebrospinal fluid (CSF) of patients with spinal cord injury. Adipose-derived mesenchymal stem cells (AD-MSCs) have been used in previous research studies at the Mayo Clinic. All subjects enrolled in this study will receive AD-MSC treatment, which is still experimental and is not approved by the U.S. Food and Drug Administration (FDA) for large scale use. However, the FDA has allowed the use of this agent in this research study.

DETAILED DESCRIPTION:
The proposed study is an open label, prospective Phase I safety and feasibility study of the intrathecal injection of autologous culture-expanded AD-MSCs in patients with severe traumatic spinal cord injury (SCI). All subjects will receive the same dosage of stem cells via intrathecal injection. Enrolled subjects will first undergo a minor surgical procedure in which a sample of the patient's adipose tissue will be harvested from a small incision in the patient's abdomen or thigh. The subject's adipose tissue will then be used to derive and culture-expand AD-MSCs for 4-6 weeks. Autologous AD-MSCs will be transplanted through intrathecal injection at the level of L4-5 under fluoroscopic guidance at a single dose of 100 million cells. Patients will be evaluated at set intervals following the injection: day 2, day 3, week 1, week 2, week 4, week 24, weeks 48, week 72 and week 96.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 years and older

   1. Females of childbearing potential must have a negative pregnancy test prior to receiving the study drug and will agree to use adequate contraception (hormonal/barrier method or abstinence) from the time of screening to a period of 1 year following completion of the drug treatment cycle. Females of childbearing potential are defined as premenopausal and not surgically sterilized, or post-menopausal for fewer than 2 years. If the urine pregnancy test is positive, the study drug will not be administered and the result will be confirmed by a serum pregnancy test. Serum pregnancy tests will be performed at a central clinical laboratory, whereas urine pregnancy tests will be performed by qualified personnel using kit.
   2. Females becoming pregnant during the study will continue to be monitored for the duration of the study or completion of the pregnancy, whichever is longer. Monitoring will include perinatal and neonatal outcome. Any SAEs associated with pregnancy will be recorded.
2. AIS grade A or B of SCI
3. SCI must be traumatic, blunt/non-penetrating in nature and not degenerative
4. SCI must be within two weeks and up to 1 year after the event
5. Full understanding of the requirements of the study and willingness to comply with the treatment plan, including fat harvesting, laboratory tests, diagnostic imaging, complete physical and neurologic examination and follow-up visits and assessments
6. Once the nature of the study is fully explained and prior to any study-related procedure is initiated the subject is willing to provide written, informed consent and complete HIPAA documentation

Exclusion Criteria:

1. Pregnant or nursing, or planning on becoming pregnant during the study period
2. AIS grade of SCI other than A or B
3. History of intra-spinal infection
4. History of superficial infection in the index spinal level within 6 months of study
5. Evidence of current superficial infection affecting the index spinal level at the time of enrollment
6. On chronic, immunosuppressive transplant therapy or having a chronic, immunosuppressive state, including use of systemic steroids/corticosteroids
7. Taking anti-rheumatic disease medication (including methotrexate or other antimetabolites) within 3 months prior to study enrollment
8. Ongoing infectious disease, including but not limited to tuberculosis, HIV, hepatitis, and syphilis
9. Fever, defined as temperature above 100.4 F/38.0 Celsius, or mental confusion at baseline
10. Significant improvement between the time of adipose tissue harvest and the time of injection, defined as improvement from AIS grade A or B to AIS grade C or greater.
11. Clinically significant cardiovascular (e.g. history of myocardial infarction, congestive heart failure or uncontrolled hypertension > 90 mmHg diastolic and/or 180 mmHg systolic), neurological (e.g. stroke, TIA) renal, hepatic or endocrine disease (e.g. diabetes, osteoporosis).
12. History of malignancy including melanoma with the exception of localized skin cancers (with no evidence of metastasis, significant invasion, or re-occurrence within three years of baseline). Any other malignancy will not be allowed.
13. History of blood dyscrasia, including but not limited to anemia, thrombocytopenia, and monoclonal gammopathy
14. Participation in a study of an experimental drug or medical device within 3 months of study enrollment
15. Known allergy to local anesthetics of other components of the study drug
16. Any contraindication to MRI scan according to MRI guidelines, or unwillingness to undergo MRI procedures
17. History of or current evidence of alcohol or drug abuse or dependence, recreational use of illicit drug or prescription medications, or use of medical marijuana within 30 days of study entry
18. Patients with baseline depression, diagnosed by the Beck Depression Inventory Assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
Incidence of acute adverse events | up to 4 weeks post treatment
  An adverse event is defined any untoward or undesirable medical occurrence in the form of signs, symptoms, abnormal findings, or diseases that emerge or worsen relative to baseline (i.e., if present upon study entry) during the study regardless of causal relationship to the study drug

SECONDARY OUTCOMES:
Incidence of delayed adverse events | 48 weeks post treatment
  An adverse event is defined any untoward or undesirable medical occurrence in the form of signs, symptoms, abnormal findings, or diseases that emerge or worsen relative to baseline (i.e., if present upon study entry) during the study regardless of causal relationship to the study drug.
Severity of adverse events | 4 weeks post-treatment
  The severity of adverse events will be graded into the following categories: mild, moderate, and severe.
Relationship of adverse events to study drug | 4 weeks post-treatment
  The relationship of adverse events to study drug will be graded into the following categories: probable, possible, unlikely, unrelated.
Incidence of serious adverse events (SAE) | 48 weeks post-treatment
  SAE is defined as adverse events that result in death, life threatening adverse experiences, hospitalization, new or prolonged disability/incapacity.
Change in sensory and motor function following completion of treatment as measured by the American Spinal Injury Association (ASIA) Impairment Scale (AIS) | baseline, 96 weeks
  The ASIA Impairment Scale describes a person's functional impairment (both motor and sensory) as a result of their spinal cord injury. The scale has 5 levels, ranging from A (complete) to E (normal).
Change in sensory and motor function following completion of treatment as measured by motor evoked potentials (MEP) | baseline, 96 weeks post-treatment
  Motor Evoked Potentials (MEP) are electrical responses recorded either from muscles, or from axons of the descending motor tract, in response to electrical or magnetic stimulation of nervous system structures that govern movement. While there are many different methods for stimulation and recording, the most common approach involves transcranial electrical stimulation of the motor pathway, using subdermal needle electrodes positioned in the scalp above primary motor cortex.
Change in sensory and motor function following completion of treatment as measured by Somatosensory Evoked Potentials (SSEPs) | baseline, 96 weeks post-treatment
  Somatosensory Evoked Potentials (SSEPs) are electrical responses recorded from the nervous system following electrical stimulation of a peripheral nerve. For example, stimulation of the median nerve at the wrist produces electrical activity that travels along the sensory pathway on its way to the brain. This activity can be recorded with electrodes positioned along that pathway.
Number of subjects who develop a new pathologic mass at the spinal cord area of injection or anywhere along the spinal cord. | approximately 96 weeks post-treatment
  Patients will undergo Magnetic Resonance Imaging of the spine and the spinal cord with and without contrast.
Change in number of red blood cells following treatment | baseline, 4 weeks post-treatment
  Blood will be drawn in order to monitor for markers of systemic inflammation. The normal range of red blood cells varies slightly between laboratories but is generally between 4.2 - 5.9 million cells/cmm. This can also be referred to as the erythrocyte count and can be expressed in international units as 4.2 - 5.9 x 10^12 cells per liter.
Change in white blood cells with differential following treatment | baseline, 4 weeks post-treatment
  Serological test - Automated white cell differential. A machine generated percentage of the different types of white blood cells, usually split into granulocytes, lymphocytes, monocytes, eosinophils, and basophils.
Change in number of platelets following treatment | baseline, 4 weeks post-treatment
  Serological test: Platelets are not complete cells, but actually fragments of cytoplasm from a cell found in the bone marrow called a megakaryocyte. Platelets play a vital role in blood clotting. Normal range varies slightly between laboratories but is in the range of 150,000 - 400,000/ cmm (150 - 400 x 10^9/liter).
Change in Serum C-Reactive Protein (CRP) | baseline, 4 weeks post-treatment
  Serological test: C-reactive protein (CRP) is produced by the liver. The level of CRP rises when there is inflammation throughout the body. It is one of a group of proteins called acute phase reactants that go up in response to inflammation. C-reactive protein is measured in milligrams of CRP per liter of blood (mg/L). Normal CRP levels are below 3.0 mg/dL.
Change in Erythrocyte Sedimentation Rate (ESR) | baseline, 4 weeks post-treatment
  Serological test. The erythrocyte sedimentation rate (ESR) is the rate at which red blood cells sediment in a period of one hour. It is a common hematology test, and is a non-specific measure of inflammation. The normal range is 0-22 mm/hr for men and 0-29 mm/hr for women.
Change in Blood Urea Nitrogen (BUN) | baseline, 4 weeks post-treatment
  Serological test - basic metabolic panel. A blood urea nitrogen (BUN) test measures the amount of nitrogen in the blood that comes from the waste product urea. Urea is made when protein is broken down in the body. Urea is made in the liver and passed out of the body in the urine. A BUN test is done to see how well the kidneys are working. Results of the blood urea nitrogen test are measured in milligrams per deciliter (mg/dL).
Change in Creatinine | baseline, 4 weeks post-treatment
  Serological test - basic metabolic panel. Creatinine is a waste product produced by muscles from the breakdown of a compound called creatine. Almost all creatinine is filtered from the blood by the kidneys and released into the urine, so blood levels are usually a good indicator of how well the kidneys are working. Results are reported in mg/dL.
Change in Sodium | baseline, 4 weeks post-treatment
  Serological test - basic metabolic panel. A sodium blood test allows the doctor to see how much sodium is in the subject's blood. It helps maintain normal blood pressure, supports the work of your nerves and muscles, and regulates your body's fluid balance. A normal sodium level is between 135 and 145 milliequivalents per liter (mEq/L) of sodium.
Change in Potassium | baseline, 4 weeks post-treatment
  Serological test - basic metabolic panel. The normal potassium level in the blood is 3.5-5.0 milliEquivalents per liter (mEq/L).
Change in Chloride | baseline, 4 weeks post-treatment
  Serological test - basic metabolic panel. The normal blood reference range of chloride for adults in most labs is 96 to 106 milliequivalents (mEq) per liter.
Change in Aspartate Aminotransferase (AST) | baseline, 4 weeks post-treatment
  Serological test - basic metabolic panel. Inflamed or injured liver cells leak higher than normal amounts of certain chemicals, including liver enzymes, into the bloodstream, which can result in elevated liver enzymes on blood tests. The reference range for aspartate aminotransferase (AST) is as follows: Males: 6-34 IU/L, Females: 8-40 IU/L.
Change in Glucose | baseline, 4 weeks post-treatment
  Serological test - basic metabolic panel. For a subject without diabetes, a fasting blood sugar on awakening should be under 100 mg/dl.
Change in Carbon Dioxide | baseline, 4 weeks post-treatment
  Serological test - basic metabolic panel. The normal range for carbon dioxide is 23 to 29 mEq/L (milliequivalent units per liter of blood).

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Bydon, MD, Principal Investigator — Mayo Clinic, Rochester, MN
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bydon M, Qu W, Moinuddin FM, Hunt CL, Garlanger KL, Reeves RK, Windebank AJ, Zhao KD, Jarrah R, Trammell BC, El Sammak S, Michalopoulos GD, Katsos K, Graepel SP, Seidel-Miller KL, Beck LA, Laughlin RS, Dietz AB. Intrathecal delivery of adipose-derived mesenchymal stem cells in traumatic spinal cord injury: Phase I trial. Nat Commun. 2024 Apr 1;15(1):2201. doi: 10.1038/s41467-024-46259-y. PMID 38561341
- [Derived] Bydon M, Dietz AB, Goncalves S, Moinuddin FM, Alvi MA, Goyal A, Yolcu Y, Hunt CL, Garlanger KL, Del Fabro AS, Reeves RK, Terzic A, Windebank AJ, Qu W. CELLTOP Clinical Trial: First Report From a Phase 1 Trial of Autologous Adipose Tissue-Derived Mesenchymal Stem Cells in the Treatment of Paralysis Due to Traumatic Spinal Cord Injury. Mayo Clin Proc. 2020 Feb;95(2):406-414. doi: 10.1016/j.mayocp.2019.10.008. Epub 2019 Nov 27. PMID 31785831
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials